CLINICAL TRIAL: NCT07400172
Title: AI-Generated Video Feedback to Improve Technical Skills in Coronary Artery Bypass Grafting
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Principal Investigator, Shengshou Hu, Prof, China National Center for Cardiovascular Diseases
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FW-HSS
Record Dates: First submitted 2025-12-23; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Cardiac; Surgery (Cardiac); Education; Artificial Intelligence (AI)
Keywords: Coronary Artery Bypass Grafting; Surgical Education; Video-Based Feedback; Artificial Intelligence

STUDY DESIGN:
Intervention Model Description: This study uses a single-group, self-controlled interventional model. Each participating cardiac surgeon acts as their own control by comparing technical skill performance before and after receiving an AI-generated targeted video feedback intervention. The intervention consists of personalized surgical video clips highlighting suboptimal technical maneuvers identified by an AI-based assessment model. No randomization or control group is involved. The study evaluates changes in surgical skill scores assessed by blinded human experts pre- and post-intervention to determine the potential educational impact of the AI feedback.
Masking Description: Human raters were blinded to surgeon identity and study phase.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AI-Guided Video Feedback Intervention (Experimental): Participants in this study will receive a personalized educational intervention consisting of AI-generated video feedback based on their baseline coronary artery bypass grafting (CABG) surgical videos. The AI model analyzes surgical performance and identifies specific operative steps with lower technical skill scores. Curated video clips highlighting these areas are provided to the surgeons for self-review and reflection. No additional formal training or coaching is given during the one-month intervention period, after which a follow-up surgical video is submitted for re-evaluation.
  Interventions: Behavioral: AI-Guided Video Feedback Intervention

INTERVENTIONS:
Behavioral: AI-Guided Video Feedback Intervention — Participants in this study will receive a personalized educational intervention consisting of AI-generated video feedback based on their baseline coronary artery bypass grafting (CABG) surgical videos. The AI model analyzes surgical performance and identifies specific operative steps with lower technical skill scores. Curated video clips highlighting these areas are provided to the surgeons for self-review and reflection. No additional formal training or coaching is given during the one-month intervention period, after which a follow-up surgical video is submitted for re-evaluation.

SUMMARY:
This study aims to evaluate whether targeted video feedback generated by an artificial intelligence (AI)-based surgical performance assessment model can support improvement in technical skills among cardiac surgeons performing coronary artery bypass grafting (CABG). This is a single-group, self-controlled, pre-post interventional study. Participating surgeons will submit a baseline CABG surgical video, which will be assessed by both an AI model and blinded human expert raters using standardized scoring criteria. Based on the AI assessment, surgeons will receive personalized video feedback highlighting operative steps associated with lower technical performance. After a one-month self-directed review period, a follow-up CABG surgical video will be submitted and evaluated using the same process. Changes in human-rated technical skill scores between baseline and follow-up will be used to assess the potential educational impact of AI-generated video feedback.

DETAILED DESCRIPTION:
Coronary artery bypass grafting (CABG) is a complex surgical procedure that requires a high level of technical skill from cardiac surgeons. Variability in surgical technique may influence procedural quality and patient outcomes. Recent advances in artificial intelligence (AI) have enabled automated assessment of surgical performance using operative video data, creating new opportunities for objective feedback and surgical education.

This study aims to evaluate whether targeted video feedback generated by an AI-based surgical performance assessment model can help cardiac surgeons improve their technical skills in CABG procedures. Participating surgeons whose baseline technical performance ranked in the lower half of the AI scoring system will receive personalized video feedback highlighting operative steps and maneuvers associated with lower performance scores.

In this single-group, self-controlled study, each participating surgeon will submit a baseline CABG surgical video, which will be independently evaluated by both the AI model and a panel of experienced cardiac surgeons using standardized scoring criteria. After receiving AI-generated video feedback, surgeons will be given one month to review and reflect on the feedback without additional formal training or coaching. A follow-up CABG surgical video will then be submitted and assessed using the same evaluation process.

The primary outcome of the study is the change in technical skill scores assigned by human expert raters between the baseline and follow-up videos. Secondary outcomes include surgeons' self-assessments of AI-identified performance deficits, agreement between AI-generated feedback and human expert feedback, and selected patient postoperative in-hospital outcomes. The findings of this study may inform the role of AI-assisted video feedback as a scalable educational tool for surgical skill development.

ELIGIBILITY:
Inclusion Criteria:

* Baseline AI-assessed technical performance ranked in the lower 50% within the scoring system in CAMERA study (NCT06739005)

Exclusion Criteria:

* Unwilling to attend

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Change in Human Expert-Rated Technical Skill Score Between Baseline and Follow-Up CABG Videos | Baseline, 1 month
  The primary outcome is the change in technical skill scores assigned by a panel of blinded human expert raters, who independently evaluate anonymized coronary artery bypass grafting (CABG) surgical videos submitted at baseline and one month after receiving AI-generated video feedback. The scoring uses a standardized rubric to assess overall surgical technical performance. The higher score, the better performance: respect for tissue, time and motion, instrument handling, knowledge of instruments, use of assistants, flow of operation and forward planning, and knowledge of the specific procedure. Each domain was scored on a 5-point Likert scale, where 1 indicated poor performance and 5 represented excellence. In addition, each rater provided an overall impression score (1-5) to capture their holistic assessment of surgical performance. The two scores were scaled to 100 points and the final score consists of 70% of 7-domain rating sum scores and 30% of overall impression score.

SECONDARY OUTCOMES:
Surgeon self-assessments of the AI feedback | 1 month
  Surgeons will review the AI-generated video clips highlighting technical performance deficits and complete a self-assessment questionnaire evaluating their satisfaction of the AI feedback.
Consistency between AI feedback and human expert feedback. | Baseline, 1 month
  This outcome assesses the consistency between the AI-generated surgical performance feedback and evaluations provided by human expert raters. AI-score was generated by a two-stage deep learning framework and human expert raters' score was generated by a validated 7-domain rating scale as detailed in the primary outcome. The intraclass correlation coefficient (ICC) will be used to assess the consistency between the surgical technique scores assessed by the AI model and those rated by human expert raters.
Postoperative in-hospital outcomes: the icidence of major complications | Baseline, 1 month
  Patient postoperative in-hospital outcomes will be collected and analyzed to explore any associations with changes in surgeon technical performance following the AI feedback intervention. The incidence of major complications (a composite outcome of death, acute kidney injury, myocardial infarction and stroke)
Postoperative in-hospital outcomes: the incidence of death | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of death.
Postoperative in-hospital outcomes: the incidence of acute kidney injury | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of acute kidney injury.
Postoperative in-hospital outcomes: the incidence of myocardial infarction | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of myocardial infarction.
Postoperative in-hospital outcomes: the incidence of stroke | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of stroke.
Postoperative in-hospital outcomes: the incidence of secondary thoracotomy | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of secondary thoracotomy.
Postoperative in-hospital outcomes: the incidence of IABP implantation | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of IABP implantation.
Postoperative in-hospital outcomes: the incidence of ECMO implantation | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of ECMO implantation.
Postoperative in-hospital outcomes: the incidence of bedside hemofiltration | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of bedside hemofiltration.
Postoperative in-hospital outcomes: the incidence of peritoneal dialysis | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of peritoneal dialysis.
Postoperative in-hospital outcomes: the incidence of tracheotomy | Baseline, 1 month
  The associations with changes in surgeon technical performance following the AI feedback intervention and the incidence of tracheotomy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Data collected for the study will be made available publicly upon reasonable request (huss@fuwai.com) after two years of publication.
Supporting Information: Study Protocol, SAP
Time Frame: After two years of publication.
Access Criteria: Anyone with a protocol sended to huss@fuwai.com and aprroved by PI can access the data. The data will be tranferred by excel or sas.